CLINICAL TRIAL: NCT07042282
Title: Comparison of Initial Treatment for Carpal Tunnel Syndrome Related to Rheumatic Diseases: Corticosteroid Injection Versus Nighttime Splinting - A Pragmatic, Open-Label, Multicenter, Randomized Clinical Trial
Brief Title: Comparison of Initial Treatment for Carpal Tunnel Syndrome Related to Rheumatic Diseases: Corticosteroid Injection Versus Nighttime Splinting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yun Qian (Other)
Collaborators: Shanghai 6th People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Yun Qian, Principal Investigator, Shanghai 6th People's Hospital
Organization: Shanghai 6th People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KY-096
Record Dates: First submitted 2025-06-25; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Carpal Tunnel Syndrome (CTS); Rheumatic Diseases
MeSH Terms: conditions — Carpal Tunnel Syndrome; Rheumatic Diseases | interventions — Adrenal Cortex Hormones; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nighttime splinting (Other): Wear a wrist neutral position splint at night for 6 weeks as the initial treatment.
  Interventions: Device: Nighttime Splinting; Other: Evaluation and Dynamic Adjustment
- Corticosteroid injection (Other): Local corticosteroid injection (triamcinolone acetonide 40mg) as the initial treatment.
  Interventions: Drug: Corticosteroid Injection; Other: Evaluation and Dynamic Adjustment

INTERVENTIONS:
Device: Nighttime Splinting — Nighttime splinting for 6 weeks.
  Other Names: Wrist Splint
  Arms: Nighttime splinting
Drug: Corticosteroid Injection — Local corticosteroid injection (triamcinolone acetonide 40mg). A single injection of triamcinolone acetonide 40mg mixed with an equal volume of 1% lidocaine is administered. The injection is performed under ultrasound guidance and anatomical landmarks to target the proximal carpal tunnel. With the wrist extended, the needle is typically inserted on the ulnar side of the palmaris longus tendon, approximately 1 cm proximal to the wrist crease. If blood is aspirated or the patient reports paresthesia (which usually indicates nerve irritation), the injection site should be adjusted.
  Other Names: Steroid Injection
  Arms: Corticosteroid injection
Other: Evaluation and Dynamic Adjustment — 6 weeks later, all patients will undergo evaluation of their initial treatment. Further therapeutic decisions will be made based on physician assessment, including: continuing nighttime splinting, administering corticosteroid injections to patients who initially received only the splint, adding nighttime splinting for patients initially received only corticosteroid injections, and transitioning from nighttime splint use to continuous wear. Subsequently, evaluations will be conducted every 6 weeks, with dynamic adjustments to the treatment plan. Throughout the study period, physicians will perform electrophysiological examinations according to changes in patients' clinical status.

SUMMARY:
The aim of this study is to evaluate the effects of corticosteroid injection verses nighttime splinting as initial treatments on wrist function, quality of life, and sleep quality in patients with rheumatoid disease-related carpal tunnel syndrome. Participants will be randomly assigned to two groups and will receive the following interventions: one group will wear a neutral position night splint for 6 weeks, and the other group will receive a single local injection of methylprednisolone 40 mg as the initial treatment. Follow-up evaluations will be conducted at 6, 12, and 18 weeks to assess wrist function, sleep quality, and quality of life, and to dynamically adjust the treatment plan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged no less than 18 years old with unilateral or bilateral carpal tunnel syndrome diagnosed by a specialist according to the Katz diagnostic criteria, and with at least one associated rheumatic disease;
2. Patients have had symptoms of CTS for at least six weeks, and the side with more severe symptoms is designated as the target side for the study.
3. During the current episode, the target side has not been treated.

Exclusion Criteria:

1. Patients who have plan for surgical treatment on his or her CTS within the following 6 months;
2. Received corticosteroid injections in the wrist within the past 6 months;
3. Patients who are unable to wear a splint due to trauma or other reasons;
4. Patients with clinical manifestations or electrophysiological changes indicative of significant axonal loss or denervation, including thenar muscle atrophy, sensory loss (two-point discrimination greater than 8 mm), absence of SNAP (sensory nerve action potential), absence of CMAP (compound muscle action potential) in the thenar muscles, etc.;
5. Patients who require long-term use of any form of opioids.
6. Patients who have used opioids (e.g., tramadol) or neuropathic pain medications (gabapentin, pregabalin, etc.) within the past 2 weeks;
7. Patients who have received non-recommended wrist injection treatments (e.g., 5% glucose, platelet-rich plasma, ozone, chitosan, hyaluronic acid, etc.) within the past 6 months;
8. Patients who have undergone non-recommended physical therapies (e.g., electrotherapy, magnetotherapy, laser therapy, etc.) within the past 6 months;
9. Patients who are pregnant or plan to become pregnant within the next 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in BCTQ function status subscale at 6 weeks | 0,6 weeks
  Change from baseline in the score of the BCTQ function status subscale (Boston Carpal Tunnel Questionnaire Function Status Subscale) will be compared between treatment groups at 6 weeks follow-up.
Change from baseline in BCTQ symptom severity subscale at 6 weeks | 0,6 weeks
  Change from baseline in the score of the BCTQ symptom severity subscale (Boston Carpal Tunnel Questionnaire Symptom Severity subscale) will be compared between treatment groups at 6 weeks follow-up.

SECONDARY OUTCOMES:
Change from baseline in BCTQ symptom severity subscale | 0,12,18 weeks
  Change from baseline in the score of the BCTQ symptom severity subscale (Boston Carpal Tunnel Questionnaire Symptom Severity subscale) will be compared between treatment groups at 12,18 weeks follow-up.
Change from baseline in BCTQ function status subscale | 0,12,18 weeks
  Change from baseline in the score of the BCTQ function status subscale (Boston Carpal Tunnel Questionnaire Function Status Subscale) will be compared between treatment groups at 12,18 weeks follow-up.
Change from baseline of EQ-VAS | 0,6,12,18 weeks
  The EQ-VAS is a measure of the overall health of respondents on the day of the survey. Change from baseline in the score of EQ-VAS will be compared between treatment groups at 6, 12, 18 weeks follow-up.
Change from baseline of PSQI | 0,6,12,18 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire that assesses sleep quality. Change from baseline in the score of the PSQI will be compared between treatment groups at 6 ,12 and 18 weeks follow-up.
Change from baseline of the cross-sectional area of the median nerve | 0,18 weeks
  The median nerve cross-sectional area will be measured with musculoskeletal ultrasound. Change from baseline of the cross-sectional area will be compared at 18 weeks follow-up.
Surgical rate within 18 weeks | 18 weeks
  Participants will be asked if they undergo surgery (carpal tunnel decompression) in the last 18 week.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Jinjiang Municipal Hospital(Shanghai Sixth People's Hospital Fujian Campus), Jinjiang, Fujian
  - Yancheng Third People's Hospital, Yancheng, Jiangsu
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study for publication, by reasonable request via email to the corresponding author.